CLINICAL TRIAL: NCT04729140
Title: A Randomized Double-blinded Placebo-controlled Outpatient Clinical Trial in High Risk Population Confirmed COVID-19 Patients Using Ivermectin and Doxycycline to Prevent COVID-19 Illness-related Hospitalization (COVIVER-OUT PLUS)
Brief Title: An Outpatient Clinical Trial Using Ivermectin and Doxycycline in COVID-19 Positive Patients at High Risk to Prevent COVID-19 Related Hospitalization
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Max Health, Subsero Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COVIVER-OUT PLUS
Record Dates: First submitted 2020-12-30; First posted 2021-01-28 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: COVID 19; Ivermectin; Doxycycline
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Doxycycline

STUDY DESIGN:
Intervention Model Description: Double-blinded, prospective, placebo controlled outpatient randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Data analysis will be carried out using statistical package for the social sciences software (SPSS). Interim data analysis will be performed at three different levels of the number of participants starting at sample size 20, 30 and 50. If no significant findings are obtained from the data at N=50, then it will add more participants to the study to achieve statistical significance. Sponsor and Principal Investigator will defer data analysis to a statistician. A Data Monitoring Committee (DMC) is going to be established in order to review accumulating trial data by treatment group in order to monitor patient safety and efficacy, ensure validity and integrity of the trial and make benefit-risk assessment. This is going to be conducted by a third party external DMC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ivermectin plus Doxycycline (Active Comparator): Ivermectin 200 mcg/kg on day 1 and day 2-plus doxycycline 100 mg tablets twice a day for seven days
  Body Weight (kg) Single oral Dose number of 3 mg tablets of Ivermectin
  15-24 kg 1 tablet
  25-35 kg 2 tablets
  36-50 kg 3 tablets
  51-65 kg 4 tablets
  66-79 kg 5 tablets
  80-109 kg 6 tablets
  >110 kg 7 tablets
  Interventions: Drug: Ivermectin Tablets; Drug: Doxycycline Tablets
- Ivermectin plus Placebo (Active Comparator): Ivermectin 200 mcg/kg on day 1 and day 2-plus placebo tablet twice a day for seven days
  Body Weight (kg) Single oral Dose number of 3 mg tablets of Ivermectin and Placebo
  15-24 kg 1 tablet
  25-35 kg 2 tablets
  36-50 kg 3 tablets
  51-65 kg 4 tablets
  66-79 kg 5 tablets
  80-109 kg 6 tablets
  >110 kg 7 tablets
  Interventions: Drug: Ivermectin Tablets; Drug: Placebo
- Placebo plus Placebo (Placebo Comparator): Placebo (number of tablets according to weight) plus placebo twice a day for seven days
  Body Weight (kg) Single oral Dose number of 3 mg tablets of Placebo
  15-24 kg 1 tablet
  25-35 kg 2 tablets
  36-50 kg 3 tablets
  51-65 kg 4 tablets
  66-79 kg 5 tablets
  80-109 kg 6 tablets
  >110 kg 7 tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin Tablets — Double-blinded, prospective, placebo controlled outpatient randomized clinical trial.
  Arms: Ivermectin plus Doxycycline; Ivermectin plus Placebo
Drug: Doxycycline Tablets — Double-blinded, prospective, placebo controlled outpatient randomized clinical trial.
  Arms: Ivermectin plus Doxycycline
Drug: Placebo — Double-blinded, prospective, placebo controlled outpatient randomized clinical trial.
  Arms: Ivermectin plus Placebo; Placebo plus Placebo

SUMMARY:
The purpose of this Clinical trial is to explore the therapeutic benefits of Ivermectin and Doxycycline in different combinations in high risk patients diagnosed with COVID-19.

DETAILED DESCRIPTION:
Purpose of the study:

The purpose of this Clinical trial is to explore the therapeutic benefits of Ivermectin and Doxycycline in different combinations. The investigators are studying known medications at already FDA approved dosages for therapeutic benefit. The investigators are not seeking new indications for these medications.

Null Hypothesis:

The investigators hypothesize that treating high-risk populations positive for COVID-19 illness with Ivermectin, Doxycycline, or Ivermectin only in the outpatient setting will decrease hospitalizations related to COVID-19 illness in comparison with Placebo.

Sample Size: Minimum of 50 high risk COVID 19 positive patients who volunteer and provide consent to participate in this study to be placed in three different groups (A,B,C). Subjects are to be randomized 1:1:1 and enrolled in sequential order to Group A, then B, then C as they enroll. This distribution pattern will be followed for the entirety of the study.

Group A: Ivermectin plus Doxycycline Group B: Ivermectin plus Placebo Group C: Placebo plus Placebo

Drug Dosing schedule:

Group A: Ivermectin 200 mcg/kg on day 1 and day 2-plus doxycycline 100 mg tablets twice a day for seven days

Group B: Ivermectin 200 mcg/kg on day 1 and day 2-plus placebo tablet twice a day for seven days

Group C: Placebo (number of tablets according to weight) plus placebo twice a day for seven days

Body Weight (kg) Table for tablets of Ivermectin

15-24 kg 1 tablet 25-35 kg 2 tablets 36-50 kg 3 tablets 51-65 kg 4 tablets 66-79 kg 5 tablets 80-109 kg 6 tablets >110 kg 7 tablets

The designated pharmacy will provide pre-packed treatment to patients based on the order of enrollment to the clinical trial.

Methods:

(A) Upon diagnosis of COVID-19 with NAAT-PCR or Rapid Antigen Test for SARS-COV 2, patients will be evaluated by their primary care physician who will consider the health risk of patients and provide all alternatives. Primary care physicians will recommend these patients to a treatment hotline number. Patients can also self refer to the treatment hot line. Patients will call this provided hotline number, and if they wish to be a part of the above said clinical trial, it will connect them to the Principal Investigator's (Dr Werther Marciales) Team. Based on inclusion and exclusion criteria, patients will be assigned to one of three different study groups outlined above. Each participant in all randomized groups will receive treatment as specified above as soon as the patient signs consent and agrees to participate in said clinical trial. Patient's subjective data including but not limited to age, gender, height, weight, detailed medical history, or any objective data will be collected and kept confidential.

(B) Patients will undergo blood work (CBC, CMP, Ferritin, D-dimer, CRP, CK, PT/INR, PTT and Fibrinogen, Interleukin 6 level,TNF alpha level, IL6 receptor level and TNF alpha receptor level) at baseline. Blood work will be repeated on days 7 and 14. These medications used in the clinical study will have a good safety profile, which has been tested over a period of time. All patients enrolled in the trial will be thoroughly evaluated prior to detailed history, especially regarding home medications, and severe co-morbid conditions as listed in the exclusion criteria.

(C) During the clinical trial, the study doctor, or the subject's primary care provider will be involved in treatment of subjects if and when there are any adverse reactions or if subjects need additional care. If a patient's COVD-19 relayed symptoms worsen then, he/she would be admitted to the hospital for further care, including mechanical ventilation if required. These patients clinical data will be followed for the remainder of he hospitalization. A patient admitted to the hospital for COVID-19 related illness will be considered to reach outcome.

Criteria for admission of confirmed COVID-19:

A patient must have COVID-19 illness and at least one of the following two conditions:

1. At least 2 of the CURB-65 criteria
2. SpO2 <93% on room air or a 4% decrease from baseline

CURB 65 criteria

1. Confusion of new onset
2. Blood Urea Nitrogen greater then 7 mmol/L (19 mg/dl)
3. Respiratory rate of 30 breaths per minute or greater
4. Blood Pressure less then 90 mm Hg systolic or 60 mm Hg diastolic
5. Age 65 or older

(D) Patients will be advised to quarantine themselves and record their temperature twice daily and maintain a home log. Patients will obtain a pulse oximeter to monitor their oxygen levels at least twice a day. Patients will also be submitted to symptoms questionnaire or ARDS questionnaire either in person or over telephone or through televist twice a week for total of five weeks.

(E) All treatment groups will also be monitored for any adverse events related to medication therapy during treatment and for 4 weeks thereafter on a twice a week basis using ADR Monitoring form. All moderate and severe adverse drug reactions will be notified to the principal investigator for immediate actions, which might include discontinuation of therapy after establishing a causal relationship. All adverse drug reactions will be recorded and reported to the FDA using Form 3500, which will be faxed to 1 800 FDA 0178. Due to the severe nature of transmissibility of COVID-19 and the importance of minimizing human interaction and preservation of Personal Protective Equipment, patients will be followed either in person, telephonically or via Televisit. Exclusion Criteria will mitigate the risk of involving patients susceptible to side effects of study treatment medications.

Data Analysis:

The total sample size is estimated at 150 participants (Minimum 50 patients in each group). The one-way analysis of variance (ANOVA) will compare group differences at baseline, midpoint, and endpoint. Data analysis will be carried out using statistical package for the social sciences software (SPSS). Interim data analysis will be performed at three different levels of the number of participants starting at sample size 20, 30 and 50. If no significant findings are obtained from the data at N=50, then it will add more participants to the study to achieve statistical significance. Sponsor and Principal Investigator will defer data analysis to a statistician. A Data Monitoring Committee (DMC) is going to be established in order to review accumulating trial data by treatment group in order to monitor patient safety and efficacy, ensure validity and integrity of the trial and make benefit-risk assessment. This is going to be conducted by a third party external DMC.

Ethical Considerations:

Informed consent will be obtained via phone, telecommunications, or in person and a copy of the consent will be sent to the subjects via postal mail, email or both. All information will be kept confidential. For research records, name, social security number, address, or phone number will not identify patients. In the event of any publication or presentation resulting from the research, no personally identifiable information will be shared. The investigators will keep the patients participation in the research study confidential to the extent permitted by law. Patient identifiers might be removed from data and, after such removal, the data could be used for future research or distributed to another investigator for future studies without additional informed consent from the subject.

Resources:

There is no funding available at this time, and the study will be self sponsored by MAX HEALTH.

Compensation:

There is no compensation offered as part of participation in this study.

Cost:

Patients will be charged for any services that are performed as part of their clinical care. Patients will not be compensated for travel or time. Patients are required to get their medication (s) used in the clinical trial from a dedicated pharmacy. Study drugs will be provided to the patients at no cost to the patient.

Removal from this study:

The patient may elect to withdraw from the study at any point. During the clinical trial, if a patients COVID-19 related symptoms worsen, then they would admitted to the hospital for further care, including mechanical ventilation if required, and the clinical data from this subset of patients will not be used for statistical consideration of this study. Still, these patients clinical data will be followed for the remainder of the hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* Willing and able to provide verbal /telephonic/Personal or computer based Informed Consent
* Experiencing symptoms of COVID-19 illness and tested positive for SARS CoV-2 with either PCR, NAAT or antigen testing
* Residents in a Nursing Home or long-term care facility
* Immunocompromised state, including solid organ transplant, HIV infection, other immune deficiency, immunosuppressant medication including systemic corticosteroids
* Chronic lung disease, including Chronic Obstructive Pulmonary Disease (COPD), moderate to severe asthma, cystic fibrosis, pulmonary fibrosis
* Cardiovascular Disease
* Cancer
* Hypertension
* Obesity (body mass index [BMI greater then or equal to 30 kg/m^2]
* Diabetes Mellitus
* Chronic Kidney Disease
* Chronic Liver Disease
* Cerebrovascular Disease
* Neurological Disorders including dementia
* Tobacco use disorders
* Hematologic disorders, including sickle cell disease and thalassemia

We are also interested in including a vital population to protect, considered essential workers who may not fit into the above inclusion criteria:

* Health care professionals and firefighters.
* Government officials or employees.
* Students and teachers.
* Law enforcement agents and personnel.
* Individuals who live with, and cannot isolate, from any of the above groups.

Exclusion Criteria:

* Participants under the age of 18
* Received any COVID vaccine within the last 30 days
* Contraindications to Ivermectin or Doxycycline
* History of Seizure Disorder or Epilepsy
* History of Myocardial Infarction or Heart Attack within the last one month
* Already receiving Ivermectin or Doxycycline for treatment of any other disease or disorder
* Allergies to Ivermectin or Doxycycline including angioedema, severe asthma, exfoliative dermatitis, Steven Jonson syndrome or psoriasis
* History of angioedema, exfoliative dermatitis, Steven Johnson syndrome, psoriasis
* Currently Pregnant or planning to conceive soon
* Breastfeeding
* History of prior Clostridium Difficile infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-12-28 (Estimated); Study Completion 2022-03-28 (Estimated)

PRIMARY OUTCOMES:
Decreased admission rate to the hospital secondary to respiratory illness related to COVID-19 | 5 weeks
  The investigators will be assessing for decreased admission rate to the hospital secondary to respiratory illness related to COVID-19. This will be assessed over the duration of 5 weeks.

SECONDARY OUTCOMES:
Decrease in total duration of symptoms secondary to respiratory illness related to COVID-19 | 5 weeks
  The investigators will be assessing for a decrease in total duration of symptoms secondary to respiratory illness related to COVID-19. This will be assessed over the duration of 5 weeks.
Assessment of White Blood Cell Count | 2 weeks
  The investigators will assess the patient's White Blood Cell Count (WBC) at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients White Blood Cell count in cells/Liter. The investigators will monitor for increases or decreases in the WBC count value throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Hemoglobin level | 2 weeks
  The investigators will assess the patient's Hemoglobin (Hgb) level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Hemoglobin count in grams/deciliter (g/dl). The investigators will monitor for increases or decreases in the Hgb value throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Hematocrit level | 2 weeks
  The investigators will assess the patient's Hematocrit (Hct) level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Hematocrit in units of percentage (%). The investigators will monitor for increases or decreases in the Hct value throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Platelet Count | 2 weeks
  The investigators will assess the patient's Platelet Count level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Platelet Count in units of platelets per microliter. The investigators will monitor for increases or decreases in the Platelet count throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Sodium level | 2 weeks
  The investigators will assess the patient's Sodium (Na) at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Sodium level in units of milliequivalents per liter (mEq/L). The investigators will monitor for increases or decreases in the Sodium level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Potassium level | 2 weeks
  The investigators will assess the patient's Potassium (K) at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Potassium level in units of milliequivalents per liter (mEq/L). The investigators will monitor for increases or decreases in the Potassium level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Chloride level | 2 weeks
  The investigators will assess the patient's Chloride (Cl) at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Chloride level in units of millimoles per liter (mmol/L). The investigators will monitor for increases or decreases in the Chloride level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Carbon Dioxide level | 2 weeks
  The investigators will assess the patient's Carbon Dioxide (C02) level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Carbon Dioxide level in units of millimoles per liter (mmol/L). The investigators will monitor for increases or decreases in the Carbon Dioxide level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Blood Urea Nitrogen level | 2 weeks
  The investigators will assess the patient's Blood Urea Nitrogen (BUN) level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Blood Urea Nitrogen level in units of milligrams per deciliter (mg/dL). The investigators will monitor for increases or decreases in the Blood Urea Nitrogen level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Creatinine level | 2 weeks
  The investigators will assess the patient's Creatinine (Crt) level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Creatinine level in units of milligrams per deciliter (mg/dL). The investigators will monitor for increases or decreases in the Creatinine level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Calcium level | 2 weeks
  The investigators will assess the patient's Calcium (Ca) level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Calcium level in units of milligrams per deciliter (mg/dL). The investigators will monitor for increases or decreases in the Calcium level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Glucose level | 2 weeks
  The investigators will assess the patient's Glucose level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Glucose level in units of milligrams per deciliter (mg/dL). The investigators will monitor for increases or decreases in the Glucose level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Total Bilirubin level | 2 weeks
  The investigators will assess the patient's Total Bilirubin (T bili) level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Total Bilirubin level in units of milligrams per deciliter (mg/dL). The investigators will monitor for increases or decreases in the Total Bilirubin level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Total Protein level | 2 weeks
  The investigators will assess the patient's Total Protein level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Total Protein level in units of grams per deciliter (g/dL). The investigators will monitor for increases or decreases in the Total Protein level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Albumin level | 2 weeks
  The investigators will assess the patient's Albumin level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Albumin level in units of grams per deciliter (g/dL). The investigators will monitor for increases or decreases in the Albumin level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Aspartate Aminotransferase level | 2 weeks
  The investigators will assess the patient's Aspartate Aminotransferase (AST) level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Aspartate Aminotransferase level in units of International Units per liter (IU/L). The investigators will monitor for increases or decreases in the Aspartate Aminotransferase level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Alanine Aminotransferase level | 2 weeks
  The investigators will assess the patient's Alanine Aminotransferase (ALT) level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Alanine Aminotransferase level in units of International Units per liter (IU/L). The investigators will monitor for increases or decreases in the Alanine Aminotransferase level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Alkaline Phosphatase level | 2 weeks
  The investigators will assess the patient's Alkaline Phosphatase (ALP) level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Alkaline Phosphatase level in units of International Units per liter (IU/L). The investigators will monitor for increases or decreases in the Alkaline Phosphatase level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Ferritin | 2 weeks
  The investigators will assess the patient's Ferritin level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Ferritin level measured in micrograms per liter (mg/L). The investigators will monitor for increases or decreases in the Ferritin level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of D-dimer | 2 weeks
  The investigators will assess the patient's D-dimer level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients D-dimer level measured in micrograms per milliliter fibrinogen equivalent units (mcg/mL FEU). The investigators will monitor for increases or decreases in the D-dimer level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Creatine Phosphokinase | 2 weeks
  The investigators will assess the patient's Creatine Phosphokinase level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Creatine Phosphokinase level measured in units per liter (U/L). The investigators will monitor for increases or decreases in the Creatine Phosphokinase level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of C-Reactive Protein | 2 weeks
  The investigators will assess the patient's C-Reactive Protein level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients C-Reactive Protein level measured in milligrams per liter (mg/L). The investigators will monitor for increases or decreases in the C-Reactive Protein level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Prothrombin Time and International Normalized Ratio | 2 weeks
  The investigators will assess the patient's Prothrombin Time and International Normalized Ratio (INR) at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Prothrombin Time measured in seconds and International Normalized Ratio measured in it's own units. The investigators will monitor for increases or decreases in the Prothrombin Time and International Normalized Ratio throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of activated Partial Thromboplastin Time | 2 weeks
  The investigators will assess the patient's activated Partial Thromboplastin Time at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients activated Partial Thromboplastin Time in seconds. The investigators will monitor for increases or decreases in the activated Partial Thromboplastin Time throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Fibrinogen Activity | 2 weeks
  The investigators will assess the patient's Fibrinogen Activity at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Fibrinogen Activity in milligrams per deciliter (mg/dl). The investigators will monitor for increases or decreases in Fibrinogen Activity throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Interleukin 6 level | 2 weeks
  The investigators will assess the patient's Interleukin 6 level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Interleukin 6 level in units of picograms per milliliter (pg/mL). The investigators will monitor for increases or decreases in the Total Interleukin 6 level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Interleukin 6 receptor level | 2 weeks
  The investigators will assess the patient's Interleukin 6 receptor level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Interleukin 6 receptor level in units of picograms per milliliter (pg/mL). The investigators will monitor for increases or decreases in the Total Interleukin 6 level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Tumor Necrosis Factor Alpha level | 2 weeks
  The investigators will assess the patient's Tumor Necrosis Factor Alpha level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Tumor Necrosis Factor Alpha level in units of picograms per milliliter (pg/mL). The investigators will monitor for increases or decreases in the Tumor Necrosis Factor Alpha level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Assessment of Tumor Necrosis Factor Alpha Receptor level | 2 weeks
  The investigators will assess the patient's Tumor Necrosis Factor Alpha Receptor level at the onset of trial enrollment and at day 7 and day 14. The investigator's will monitor the patients Tumor Necrosis Factor Alpha Receptor level in units of picograms per milliliter (pg/mL). The investigators will monitor for increases or decreases in the Tumor Necrosis Factor Alpha Receptor level throughout the first 2 weeks of trial enrollment. Participants will have their blood work sent to a designated laboratory.
Mortality | 5 weeks
  The investigators will assess for any reductions or increase in mortality during the duration of the study.
Measurement of Participants with Medication Side Effects | 5 weeks
  The investigators will assess for new onset of medication side effects on a twice a week basis for the duration of 5 weeks using a standardized form. The investigators will ask about rash/itching/hives, bleeding/easy bruising of skin, palpitations or irregular heart beats, vision disturbances or blurry vision, light flashes or light streak in vision, fainting spells, seizure, headaches, nausea or vomiting, ringing in the ears, loss of appetite, loss of taste sensation, oral ulcers, abdominal pain, diarrhea or loss stools, yellow discoloration of eyes or skin, upper extremity or lower extremity muscle weakness, mood changes, teeth discoloration, photosensitivity or sunburn reactions after sun exposure, or any other effects. This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Shortness of Breath or Changes in Shortness of Breath Severity | 5 weeks
  The investigators will assess for new onset Shortness of Breath or changes in the severity of Shortness of Breath on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if Shortness of Breath is present and grade the severity of Shortness of Breath if present (mild, moderate, severe). Moderate to Severe Shortness of Breath will be immediately reported to the Principal Investigator. This may occur via Tele-Health visits or via in person visits.
Measurement of Participants Pulse Oximetry readings on room air | 5 weeks
  The investigators will assess Pulse Oximetry readings on room air on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record Pulse Oximetry readings on room air. If the Pulse Oximetry readings on room air are less then 93% on room air or drop by 4% from baseline established at the onset of the study, the Prinicipal Investigator will be notified. This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Red Eyes or Changes in Red Eyes Severity | 5 weeks
  The investigators will assess for new onset of Red Eyes or changes in the severity of Red Eyes on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if Red Eyes are present and grade the severity of Red Eyes if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Chills or Changes in Chills Severity | 5 weeks
  The investigators will assess for new onset of Chills or changes in the severity of Chills on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if Chills are present and grade the severity of Chills if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Runny Nose or Changes in Runny Nose Severity | 5 weeks
  The investigators will assess for new onset of Runny Nose or changes in the severity of Runny Nose on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if Runny Nose is present and grade the severity of Runny Nose if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Sore Throat or Changes in Sore Throat Severity | 5 weeks
  The investigators will assess for new onset of Sore Throat or changes in the severity of Sore Throat on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if Sore Throat is present and grade the severity of Sore Throat if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Loss of Smell or Changes in Severity of in Loss of Smell | 5 weeks
  The investigators will assess for new onset of Loss of Smell or changes in the severity of Loss of Smell on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if Loss of Smell is present and grade the severity of Loss of Smell if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Loss of Taste or Changes in Severity of Loss of Taste | 5 weeks
  The investigators will assess for new onset of Loss of Taste or changes in the severity of Loss of Taste on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if Loss of Taste is present and grade the severity of Loss of Taste if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Body Aches or Body Pains or Changes in Body Aches or Body Pains Severity | 5 weeks
  The investigators will assess for new onset of Body Aches or Body Pains or changes in the severity of Body Aches or Body Pains on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if Body Aches or Body Pains are present and grade the severity of Body Aches or Body Pains if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Diarrhea or Changes in Diarrhea Severity | 5 weeks
  The investigators will assess for new onset of Diarrhea or changes in the severity of Diarrhea on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if Diarrhea is present and grade the severity of Diarrhea if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Headaches or Changes in Headaches Severity | 5 weeks
  The investigators will assess for new onset of Headaches or changes in the severity of Headaches on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if Headaches are present and grade the severity of Headaches if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Anxiety or Changes in Anxiety Severity | 5 weeks
  The investigators will assess for new onset of Anxiety or changes in the severity of Anxiety on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if Anxiety is present and grade the severity of Anxiety if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Fatigue or Changes in Fatigue Severity | 5 weeks
  The investigators will assess for new onset of fatigue or changes in the severity of fatigue on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if fatigue is present and grade the severity of fatigue if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Trouble Concentrating or Changes in Trouble Concentrating Severity | 5 weeks
  The investigators will assess for new onset of Trouble Concentrating or changes in the severity of Trouble Concentrating on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if Trouble Concentrating is present and grade the severity of Trouble Concentrating if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Cough or Changes in Cough Severity | 5 weeks
  The investigators will assess for new onset of cough or changes in the severity of cough on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if cough is present and grade the severity of cough if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Vomiting or Changes in Vomiting Severity | 5 weeks
  The investigators will assess for new onset of vomiting or changes in the severity of vomiting on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if vomiting is present and grade the severity of vomiting if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Nausea or Changes in Nausea Severity | 5 weeks
  The investigators will assess for new onset of nausea or changes in the severity of nausea on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if nausea is present and grade the severity of nausea if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Feelings of Hopelessness or Changes in Feelings of Hopelessness severity | 5 weeks
  The investigators will assess for new onset of feelings of hopelessness or changes in the severity of feelings of hopelessness on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if feelings of hopelessness are present and grade the severity of hopelessness if present (mild, moderate, severe). If more then mild, the investigators will utilize the Hamilton Depression Scale. This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset feelings of Depression or Changes in feelings of Depression severity | 5 weeks
  The investigators will assess for new onset of feelings of depression or changes in the severity of feelings of depression on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if feelings of depression are present and grade the severity of feelings of depression if present (mild, moderate, severe). If more then mild, the investigators will utilize the Hamilton Depression Scale. This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Fever or Changes in Fever Severity | 5 weeks
  The investigators will assess for new onset of a fever or changes in the severity of fever on a twice a week basis for the duration of 5 weeks. The investigators will be monitoring for fever in Fahrenheit (F). The investigators will be using a standardized form which will record if fever is present and grade the severity of fever if present (mild fever at 100.4 degrees F to 101 degrees F, moderate fever at 101.1 to 101.9 degrees, severe fever at greater then 102 degrees). We will also record the temperatures in the standardized form. This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Moving Slowly or Changes in the Severity of Moving Slowly | 5 weeks
  The investigators will assess for new onset of moving slowly or changes in severity of moving slowly on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if moving slowly is present and grade the severity of moving slowly if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Speaking Slowly or Changes in the Severity of Speaking Slowly | 5 weeks
  The investigators will assess for new onset of speaking slowly or changes in severity of speaking slowly on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if speaking slowly is present and grade the severity of speaking slowly if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Feelings of Restlessness or Changes in the Severity of Feelings of Restlessness | 5 weeks
  The investigators will assess for new onset feelings of restlessness or changes in severity of feelings of restlessness on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if feelings of restlessness are present and grade the severity of these feelings of restlessness if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Thoughts of Better Off Being Dead or Changes in the Severity of Thoughts of Better Off Being Dead | 5 weeks
  The investigators will assess for new onset thoughts of better off being dead or changes in severity of thoughts of better off being dead on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if thoughts of better off being dead are present and grade the severity of these thoughts of better off being dead if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Thoughts of Hurting Yourself or Changes in the Severity of Thoughts of Hurting Yourself | 5 weeks
  The investigators will assess for new onset thoughts of hurting yourself or changes in severity of thoughts of hurting yourself on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if thoughts of hurting yourself are present and grade the severity of these thoughts of hurting yourself if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Loss of Interest in Doing Things or Changes in the Severity of Loss of Interest in Doing Things | 5 weeks
  The investigators will assess for new onset loss of interest in doing things or changes in the severity of loss of interest in doing things on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if loss of interest in doing things are present and grade the severity of the loss of interest in doing things if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Loss of Pleasure in Doing Things or Changes in the Severity of Loss of Pleasure in Doing Things | 5 weeks
  The investigators will assess for new onset loss of pleasure in doing things or changes in the severity of loss of pleasure in doing things on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if loss of pleasure in doing things are present and grade the severity of the loss of pleasure in doing things if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Trouble Falling Asleep or Changes in the Severity of Trouble Falling Asleep | 5 weeks
  The investigators will assess for new onset trouble falling asleep or changes in the severity of trouble falling asleep on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if trouble falling asleep are present and grade the severity of the trouble falling asleep if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Trouble Staying Asleep or Changes in the Severity of Trouble Staying Asleep | 5 weeks
  The investigators will assess for new onset trouble staying asleep or changes in the severity of trouble staying asleep on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if trouble staying asleep is present and grade the severity of trouble staying asleep if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.
Measurement of Participants with new onset Unmentioned Negative Impacts of COVID 19 infection or Changes in the Severity of these Negative Impacts of COVID 19 infection | 5 weeks
  The investigators will assess for new onset unmentioned negative impacts of COVID 19 infection or changes in the severity of these unmentioned negative impacts of COVID 19 infection on a twice a week basis for the duration of 5 weeks. The investigators will be using a standardized form which will record if unmentioned negative impacts of COVID 19 infection are present and grade the severity of these unmentioned negative impacts of COVID 19 infection if present (mild, moderate, severe). This may occur via Tele-Health visits or via in person visits.

CONTACTS AND LOCATIONS:
Overall Officials: Werther Marciales, MD, Principal Investigator — Clinical Trial Principal Investigator; Ryan Salom, Principal Investigator — sub Clinical Trial Prinicipal Investigator; Faheem Ahmad, MD, Principal Investigator — sub Clinical Trial Prinicipal Investigator; Divisha Sharma, MD, Principal Investigator — Clinical Trial Investigator; Nicholas Guy Ross, DO, Principal Investigator — Clinical Trial Investigator; Terry Fredeking, Principal Investigator — Clinical Trial Investogator; Michael Ricciardi, PhD, Principal Investigator — Clinical Trial Investogator
Locations (1):
- MAX HEALTH, Subsero Health 2055 Wood Street, Suite 100, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
We will release data once the clinical trial has completed course. An independent data safety committee will analyze interim data for effectiveness and safety.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: December 28 2020 to March 28 2022

REFERENCES:
- [Background] [1] World Health Organization. Novel Coronavirus-China [cited 2020 January 12]. https://www.who.int/csr/don/12-january-2020-novel-coronavirus-chinaExternal Link
- [Background] [2] Interim U.S. Guidance for Risk Assessment and Public Health Management of Persons with Potential Coronavirus Disease 2019 (COVID-19) Exposures: Geographic Risk and Contacts of Laboratory-confirmed Cases. www.cdc.gov/coronavirus/2019-ncov/php/risk-assessment.
- [Background] Holshue ML, DeBolt C, Lindquist S, Lofy KH, Wiesman J, Bruce H, Spitters C, Ericson K, Wilkerson S, Tural A, Diaz G, Cohn A, Fox L, Patel A, Gerber SI, Kim L, Tong S, Lu X, Lindstrom S, Pallansch MA, Weldon WC, Biggs HM, Uyeki TM, Pillai SK; Washington State 2019-nCoV Case Investigation Team. First Case of 2019 Novel Coronavirus in the United States. N Engl J Med. 2020 Mar 5;382(10):929-936. doi: 10.1056/NEJMoa2001191. Epub 2020 Jan 31. PMID 32004427
- [Background] Fauci AS, Lane HC, Redfield RR. Covid-19 - Navigating the Uncharted. N Engl J Med. 2020 Mar 26;382(13):1268-1269. doi: 10.1056/NEJMe2002387. Epub 2020 Feb 28. No abstract available. PMID 32109011
- [Background] [5] The RECOVERY trial in COVID-19 has provided initial results of the dexamethasone arm https://www.recoverytrial.net/files/recovery_dexamethasone_statement_160620_final.pdf
- [Background] [6] U.S. Food and Drug Administration. FDA cautions against the use of hydroxychloroquine or chloroquine for COVID-19 outside of the hospital setting or a clinical trial due to the risk of heart rhythm problems. Available at: https://www.fda.gov/drugs/drug-safety-and-availability/fda-cautions-against-use-hydroxychloroquine-or-chloroquine-covid-19-outside-hospital-setting-or (Accessed on April 24, 2020).
- [Background] [7] Georgi Momekov & Denitsa Momekova (2020) Ivermectin as a potential COVID-19 treatment from the pharmacokinetic point of view: antiviral levels are not likely attainable with known dosing regimens, Biotechnology & Biotechnological Equipment, 34:1, 469-474, DOI: 10.1080/13102818.2020.1775118
- [Background] [8] ICON (Ivermectin in COvid Nineteen) study: Use of Ivermectin is Associated with Lower Mortality in Hospitalized Patients with COVID19 Juliana CepelowiczRajter, M.D. 1 Michael S. Sherman, M.D.2NaazFatteh, M.D. 1 Fabio Vogel, Pharm. D., BCPS1 Jamie Sacks, Pharm. D. 1 Jean-Jacques Rajter, M.D.1,3 1. Broward Health Medical Center, Fort Lauderdale, FL 2. Emeritus Professor, Drexel University College of Medicine 3. Assistant Professor, Florida International University Corresponding author: Jean-Jacques Rajter, MD covid19@pscflorida.com
- [Background] [9] The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro, Leon Calya, Julian D. Drucea, Mike G. Cattona, David A. Jans, Kylie M. Wagstaffb,∗ a Victorian Infectious Diseases Reference Laboratory, Royal Melbourne Hospital, At the Peter Doherty Institute for Infection and Immunity, Victoria, 3000, Australia b Biomedicine Discovery Institute, Monash University, Clayton, Vic, 3800,
- [Background] [10] Ivermectin: a potential candidate for the treatment of COVID 19 Dhyuti Gupta 1, Ajaya Kumar Sahoo 1, Alok Singh ∗,1 Department of Pharmacology, All India Institute of Medical Sciences, Raipur, Chhattisgarh, India
- [Background] [11] Loukas A, Hotez PJ. Chemotherapy of helminth infections. In: Brunton LL, Lazo JS, Parker KL, editors. Goodman & Gilman's The pharmacological basis of therapeutics. 11th ed. New York (N.Y.): McGraw Hill; 2006. p. 1073-1093.
- [Background] Guzzo CA, Furtek CI, Porras AG, Chen C, Tipping R, Clineschmidt CM, Sciberras DG, Hsieh JY, Lasseter KC. Safety, tolerability, and pharmacokinetics of escalating high doses of ivermectin in healthy adult subjects. J Clin Pharmacol. 2002 Oct;42(10):1122-33. doi: 10.1177/009127002401382731. PMID 12362927
- [Background] Navarro M, Camprubi D, Requena-Mendez A, Buonfrate D, Giorli G, Kamgno J, Gardon J, Boussinesq M, Munoz J, Krolewiecki A. Safety of high-dose ivermectin: a systematic review and meta-analysis. J Antimicrob Chemother. 2020 Apr 1;75(4):827-834. doi: 10.1093/jac/dkz524. PMID 31960060
- [Background] [14] Dalvi P.S.; Singh A; Trivedi HR; et al. (2011).
- [Background] McCullough PA, Kelly RJ, Ruocco G, Lerma E, Tumlin J, Wheelan KR, Katz N, Lepor NE, Vijay K, Carter H, Singh B, McCullough SP, Bhambi BK, Palazzuoli A, De Ferrari GM, Milligan GP, Safder T, Tecson KM, Wang DD, McKinnon JE, O'Neill WW, Zervos M, Risch HA. Pathophysiological Basis and Rationale for Early Outpatient Treatment of SARS-CoV-2 (COVID-19) Infection. Am J Med. 2021 Jan;134(1):16-22. doi: 10.1016/j.amjmed.2020.07.003. Epub 2020 Aug 7. PMID 32771461
- [Background] [16] Goodman and Gilman's The Pharmacological Basis of Therapeutics, 11th edition, page 122, 1084-1087.
- [Background] [17] COMFORTIS® and ivermectin interaction Safety Warning Notification
- [Background] Smith K, Leyden JJ. Safety of doxycycline and minocycline: a systematic review. Clin Ther. 2005 Sep;27(9):1329-42. doi: 10.1016/j.clinthera.2005.09.005. PMID 16291409
- [Background] [19] Information for Clinicians on Therapeutic Options for COVID-19 Patients. www.cdc.gov/coronavirus/2019-ncov/hcp/therapeutic-options.
- [Background] Teuwen LA, Geldhof V, Pasut A, Carmeliet P. COVID-19: the vasculature unleashed. Nat Rev Immunol. 2020 Jul;20(7):389-391. doi: 10.1038/s41577-020-0343-0. PMID 32439870
- [Background] Sodhi M, Etminan M. Therapeutic Potential for Tetracyclines in the Treatment of COVID-19. Pharmacotherapy. 2020 May;40(5):487-488. doi: 10.1002/phar.2395. Epub 2020 May 4. No abstract available. PMID 32267566
- [Background] Henehan M, Montuno M, De Benedetto A. Doxycycline as an anti-inflammatory agent: updates in dermatology. J Eur Acad Dermatol Venereol. 2017 Nov;31(11):1800-1808. doi: 10.1111/jdv.14345. Epub 2017 Jun 7. PMID 28516469
- [Background] Yoshikawa T, Hill T, Li K, Peters CJ, Tseng CT. Severe acute respiratory syndrome (SARS) coronavirus-induced lung epithelial cytokines exacerbate SARS pathogenesis by modulating intrinsic functions of monocyte-derived macrophages and dendritic cells. J Virol. 2009 Apr;83(7):3039-48. doi: 10.1128/JVI.01792-08. Epub 2008 Nov 12. PMID 19004938
- [Background] Kritas SK, Ronconi G, Caraffa A, Gallenga CE, Ross R, Conti P. Mast cells contribute to coronavirus-induced inflammation: new anti-inflammatory strategy. J Biol Regul Homeost Agents. 2020 January-February,;34(1):9-14. doi: 10.23812/20-Editorial-Kritas. PMID 32013309
- [Background] Dutta K, Basu A. Use of minocycline in viral infections. Indian J Med Res. 2011 May;133(5):467-70. PMID 21623029
- [Background] Zakeri B, Wright GD. Chemical biology of tetracycline antibiotics. Biochem Cell Biol. 2008 Apr;86(2):124-36. doi: 10.1139/O08-002. PMID 18443626
- [Background] Phillips JM, Gallagher T, Weiss SR. Neurovirulent Murine Coronavirus JHM.SD Uses Cellular Zinc Metalloproteases for Virus Entry and Cell-Cell Fusion. J Virol. 2017 Mar 29;91(8):e01564-16. doi: 10.1128/JVI.01564-16. Print 2017 Apr 15. PMID 28148786
- [Background] Rothan HA, Mohamed Z, Paydar M, Rahman NA, Yusof R. Inhibitory effect of doxycycline against dengue virus replication in vitro. Arch Virol. 2014 Apr;159(4):711-8. doi: 10.1007/s00705-013-1880-7. Epub 2013 Oct 19. PMID 24142271
- [Background] Sargiacomo C, Sotgia F, Lisanti MP. COVID-19 and chronological aging: senolytics and other anti-aging drugs for the treatment or prevention of corona virus infection? Aging (Albany NY). 2020 Mar 30;12(8):6511-6517. doi: 10.18632/aging.103001. Epub 2020 Mar 30. PMID 32229706
- [Background] [30] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, et al. (May 2020).